CLINICAL TRIAL: NCT03630991
Title: Monitoring, Detoxifying, and Rebalancing Metals During Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS) Therapy
Brief Title: Edetate Calcium Disodium or Succimer in Treating Patients With Acute Myeloid Leukemia or Myelodysplastic Syndrome Undergoing Chemotherapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0752; NCI-2018-01610 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0752 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; High Risk Myelodysplastic Syndrome; Myelodysplastic Syndrome; Myelodysplastic/Myeloproliferative Neoplasm; Myeloproliferative Neoplasm; Recurrent Acute Myeloid Leukemia; Recurrent Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Recurrent Myelodysplastic Syndrome; Recurrent Myelodysplastic/Myeloproliferative Neoplasm; Refractory Acute Myeloid Leukemia; Refractory Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Refractory Myelodysplastic Syndrome; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndrome; Very High Risk Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Myeloproliferative Disorders | interventions — Pentetic Acid; Edetic Acid; Geritol; Succimer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort I (edetate calcium disodium, multivitamin) (Experimental): During standard of care chemotherapy, patients receive edetate calcium disodium IV daily over 30 minutes for 4 doses for each cycle. Treatment continues for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive up to 12 multivitamin capsules PO daily while on study.
  DOSE EXPANSION: During standard of care chemotherapy, patients receive edetate calcium disodium IV daily over 30 minutes for 4 doses for each cycle. DMSA daily for 21 days. Multivitamin capsules daily while on study. Patients will receive treatment for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Edetate Calcium Disodium; Dietary Supplement: Multivitamin
- Cohort II (succimer, multivitamin) (Experimental): During standard of care chemotherapy, patients receive succimer PO daily for 8 or 21 days of each cycle beginning day 1. Treatment continues for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive up to 12 multivitamin capsules PO daily while on study.
  DOSE EXPANSION: During standard of care chemotherapy, patients receive edetate calcium disodium IV daily over 30 minutes for 4 doses for each cycle. DMSA daily for 21 days. Multivitamin capsules daily while on study. Patients will receive treatment for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: Multivitamin; Drug: Succimer

INTERVENTIONS:
Drug: Edetate Calcium Disodium — Given IV
  Other Names: C10H12CaN2Na2O8; Calcium disodium edetate; Calcium Disodium Ethylenediaminetetraacetate; Calcium Disodium Versenate; Calcium EDTA; Disodium calcium ethylenediaminetetraacetate; EDTA Calcium
  Arms: Cohort I (edetate calcium disodium, multivitamin)
Dietary Supplement: Multivitamin — Given PO
  Other Names: Geritol; Vitamin Supplements (NOS)
Drug: Succimer — Given PO
  Other Names: Chemet; DMSA; Meso 2, 3-Dimercaptosuccinic Acid
  Arms: Cohort II (succimer, multivitamin)

SUMMARY:
This phase I trial studies the side effects and best dose of edetate calcium disodium or succimer in treating patients with acute myeloid leukemia or myelodysplastic syndrome undergoing chemotherapy. Edetate calcium disodium or succimer may help to lower the level of metals found in the bone marrow and blood and may help to control the disease and/or improve response to chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To establish the maximal tolerated dose (MTD) of Phase 1 in acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) patients undergoing therapy combined with succimer (DMSA) and edetate calcium disodium (Ca-EDTA). (Phase I dose escalation)
2. To assess the efficacy information regarding the combined therapy in terms of the overall response rate (ORR) including complete remission (CR), CR with partial hematological recovery (CRh), CR with incomplete count recovery (CRi), morphologic leukemia free state (MLFS), and partial remission (PR). (Phase I expansion)

SECONDARY OBJECTIVES:

1. To assess the complete remission (CR), complete remission with incomplete hematologic recovery (CRi), complete remission with partial hematological recovery (CRh), partial remission (PR), hematologic improvement (HI), morphologic leukemia free state (MLFS) rates, cytogenetic response, and the 1-year overall survival (OS) in AML patients and the CR/marrow CR/hematologic improvement (HI) rate, partial remission (PR) rate and 1-year overall survival (OS) and cytogenetic response in MDS patients undergoing MDS/AML therapy combined with DMSA and Ca-EDTA.
2. To assess overall survival and event free survival in AML and MDS patients undergoing AML and MDS therapy combined with DMSA and Ca-EDTA
3. To assess remission duration in AML and MDS patients undergoing AML and MDS therapy combined with DMSA and Ca-EDTA.
4. To monitor toxic and essential metal levels during AML and MDS therapy combined with DMSA and Ca-EDTA and to evaluate the reduction in metals in the bone marrow and blood of newly diagnosed AML and MDS patients undergoing metal detoxification combined with standard AML/MDS therapy.
5. To evaluate the safety profile in AML and MDS patients undergoing AML and MDS therapy combined with DMSA and Ca-EDTA.
6. Correlate metal and copper isotopic abundance ratios of AML and MDS patients with clinical data, conventional cytogenetics, extensive next generation sequencing (NGS) (300-gene panel), exposure survey data, and clinical outcome data, and to perform a larger analysis by pooling this data with metal/genomic/survey/outcome data obtained on 2017-0937 and PA15-0302.
7. Estimate the progression rate in MDS patients.
8. To assess other responses of interest.
9. To compare overall survival and response in this study with historical data of patients who were treated without Ca-EDTA and DMSA.

EXPLORATORY OBJECTIVES:

1. To correlate the degree of metal chelation with the degree of therapeutic response and minimal residual disease (MRD).
2. To collect environmental exposure data on the environmental health assessment survey.
3. To assess P53 folding or p53 activity before and after the first dose of Ca-EDTA chelation in MDS and AML patients, and patients with other malignancies.
4. To study changes in cytogenetic/molecular data during treatment, as well as, protein expression data (by immunohistochemistry or proteomics), including for transcription factors/tumor suppressors (e.g. TP53 and MYC).
5. To perform pre-clinical proof of concept studies of metals and metal chelators in a variety of AML cells and cell lines including: AML cell lines, primary hematologic malignancy cells, stromal cell lines, and patient-derived stromal cells.
6. To explore metal chelation in pediatric, adolescent, and young adult cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form participants ≥18 years, unless parent or LAR signs along with any required verbal assents and signed assent of minor for participants <18 years.
* Age ≥18 years at the time of signing the informed consent form.
* Age ≥1 years and <18 years with weight requirement ≥8 kg at the time of the signing of the informed consent form (e.g. by parent or LAR)
* Patients enrolling in the pediatric/adolescent/young adult exploratory cohort must be:

Age ≥1 years and <18 years with weight requirement ≥8 kg at the time of the signing of the informed consent form (e.g. by parent or LAR), Or age 18 years -39 years at the time of the signing of the informed consent form

* Diagnosis of any of the following:
* Newly diagnosed (or untreated) AML with intermediate-risk/poor-risk cytogenetics, intermediate-risk/poor-risk molecular, or secondary AML (i.e. therapy-related or evolved from antecedent hematologic malignancy)
* Newly diagnosed (or untreated) myeloid blast phase of myeloproliferative neoplasm (MPN) (including myeloid blast phase of chronic myeloid leukemia [CML])
* Newly diagnosed (or untreated) high-risk, very-high risk or secondary MDS/myeloid neoplasm
* Newly diagnosed (or untreated) MDS/MPN (regardless of cytogenetic/molecular status)
* Relapsed and/or refractory AML, MDS/myeloid neoplasm , MDS/MPN, myeloid blast phase of MPN (including myeloid blast phase of CML)
* Patients enrolling in the childhood/adolescent/young adult exploratory cohort may have any of the following diagnoses:
* High-risk or relapsed/refractory childhood, adolescent, or young adult malignancies including but not limited to high-risk or relapsed/refractory ALL or other high-risk or relapsed refractory malignancies
* This includes, but is not limited to, the following: High-risk ALL/LL including T-ALL/LL, Ph-like ALL/LL, Ph+ B-ALL/LL, B-ALL/LL with CNS lymphoid leukemic involvement, testicular involvement, other extramedullary involvement by ALL/LL; ALL/LL with any of the NCI high-risk features: patients aged 10 years or older and those with a white blood cell count ≥50 × 109 per L), high-risk cytogenetics (MLL rearrangements, near haploidy [<30 chromosomes], low hypodiploidy [30-39 chromosomes], t[17;19][q23;p13], intrachromosomal amplification of chromosome 21), Burkitts'; Burkitt's-like, Double-Hitt; CNS involvement by any non-primary brain malignancy; Metastatic disease of any malignancy; 5-year survival prognosis of less than 50%, based on the treating physician's assessment
* Patients on non-investigational regimens or on IND-exempt MD Anderson studies (for hematologic malignancies) of approved drugs are also eligible.
* Patients on IND studies (for hematologic malignancies) utilizing FDA approved commercially available drugs are eligible.
* Investigational agents that are not used for treatment of the leukemia per se (e.g. anti-infective prophylaxis or therapy) will be allowed. Other supportive care studies are allowed, even if under an IND.
* Newly diagnosed MDS or AML, as well as MDS/MPN, myeloid blast phase of MPN (including myeloid blast phase of CML), patients can enroll on this study after start of non-investigational induction therapy, but must be within first 3 cycles of therapy of front-line therapy. Patients with relapsed and/or refractory AML, MDS, MDS/MPN, myeloid blast phase of MPN (including myeloid blast phase of CML) can enroll. Newly diagnosed patients enrolling in the exploratory cohort with high-risk malignancies can enroll after the start of non-investigational therapy but must be within first 3 cycles of front-line therapy.
* Transformed and untreated AML transformed from previously treated MDS, myeloproliferative neoplasm (MPN) or other types of secondary AML are allowed. Myeloid-Blast Phase of MPN and Chronic Myeloid Leukemia (CML) are allowed.
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 3 or Lansky or Karnofsky ≥ 30 at study entry; patients who are unable to walk, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Laboratory test results within these ranges (unless due to leukemia or other hematologic malignancy):
* Serum creatinine =< 1.5 mg/dL
* Total Bilirubin =< 2.0 x upper limit of normal (ULN), unless the patient has Gilbert's
* AST (SGOT) and/or ALT (SGPT) =< 2.0 x ULN
* Women of childbearing potential (WCBP) must have a negative urine pregnancy test within 7 days and must either commit to continued abstinence from heterosexual intercourse or adopting at least one highly effective method of contraception. These methods include intra-uterine device, tubal ligation, partner's vasectomy, and hormonal birth control pills. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential
* Extramedullary disease is allowed as long as it can be measured and followed for response.

Note: Patients can be considered MDS by either WHO or FAB150 criteria Note: MDS risk status assessment is based on IPSS-R and/or IPSS-M. AML risk status assessment is based on ELN and World Health Organization classification

Exclusion Criteria:

* Nursing and pregnant females. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Uncontrolled inter-current illness including, but not limited to, uncontrolled active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements or which judged by the investigator, places the patient at unacceptable risk
* Acute Promyelocytic leukemia (APL)

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2018-10-11 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | At 30 days post-treatment
  Safety data of the patients will be summarized using descriptive statistics such as mean, standard deviation, median and range. Will follow standard reporting guidelines for adverse events. Safety data will be summarized by category, severity and frequency.
Maximum tolerated doses (MTD) of edetate calcium disodium (Ca-EDTA) and succimer (DMSA) (Phase 1 dose escalation) | Up to the end of cycle 1 (each cycle is 28 days)
  The MTD is the highest dose level in which < 2 patients of 6 develop first cycle dose-limiting toxicity (DLT).

CONTACTS AND LOCATIONS:
Overall Officials: Maro Ohanian, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org